CLINICAL TRIAL: NCT07161882
Title: Observational Study of the Epidemiological, Clinical, and Diagnostic Profile, Treatment Patterns, and Outcomes of Lung Cancer.
Brief Title: ALG-LungCancerRegistry (SAFRO2202)
Acronym: SAFRO2202
Status: Recruiting | Type: Observational
Sponsor: Société Algérienne de Formation et de Recherche en Oncologie (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 013/SAF/OBS/EPD/2024; SAFRO 2202 (Registry Identifier: ALG Lung Cancer Registry)
Record Dates: First submitted 2025-06-25; First posted 2025-09-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell; Carcinoid Tumor
Keywords: Lung Cancer; Non-Small Cell Lung Cancer; Carcinoid Tumor; Treatment Outcomes; Drug-Related Side Effects; Registries; Algeria
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell; Carcinoid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung Cancer Patients Cohort: Adult patients (≥18 years) diagnosed with lung cancer (NSCLC, SCLC, or carcinoid tumors) at the time of inclusion or within the previous 12 months, fully managed in oncology or pulmonology departments at one of the 21 participating public or university hospitals across Algeria. Data are collected prospectively during routine clinical care.
  Interventions: Other: Observational Data Collection

INTERVENTIONS:
Other: Observational Data Collection — Collection of clinical, pathological, molecular, and treatment-related data during routine care, with no additional procedures or interventions required by the study.

SUMMARY:
SAFRO 2202 ALG-Lung Cancer Registry is a prospective, multicenter, non-interventional observational study conducted across 21 public and university hospitals in Algeria. The objective is to characterize the epidemiological, clinical, pathological, molecular, and therapeutic features of patients diagnosed with lung cancer, including non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), and carcinoid tumors.

Eligible participants are adults aged 18 years or older, diagnosed at the time of inclusion or within the previous 12 months, and fully managed in oncology or pulmonology departments. Data are collected during routine clinical care and recorded in a secure electronic case report form (eCRF). No protocol-mandated interventions or study-specific visits are required.

The study plans to enroll approximately 1,500 patients per year over a 30-month period. Primary outcomes include demographic and clinical profiles, tumor histology, molecular markers, staging at diagnosis, and treatment strategies (surgery, radiotherapy, chemotherapy, targeted therapy, and immunotherapy). Secondary outcomes include treatment-related toxicities, objective response rate (ORR), progression-free survival (PFS), time to treatment discontinuation (TTD), and overall survival (OS).

The findings from this registry will provide real-world evidence to support national health planning, improve lung cancer management, and guide future clinical and public health initiatives in Algeria.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related morbidity and mortality worldwide, and its incidence continues to rise in Algeria. Despite this increasing burden, real-world data regarding the epidemiology, clinical management, and treatment outcomes of lung cancer remain limited at the national level. The SAFRO 2202 ALG-Lung Cancer Registry was established to fill this gap by systematically collecting prospective, real-life data from a large sample of patients managed within Algeria's public healthcare system.

This study is a prospective, multicenter, non-interventional observational registry conducted across 21 hospital centers specialized in oncology and pulmonology. It includes adult patients (aged ≥18 years) with a confirmed diagnosis of lung cancer, including non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), and carcinoid tumors. The study includes all patients diagnosed at the time of inclusion or within the 12 months preceding inclusion, provided they meet the eligibility criteria. All patients must be fully managed within the public healthcare system, including diagnosis, treatment, and follow-up.

Data will be collected as part of routine medical care, with no study-specific visits required, and will be entered into a secure electronic case report form (eCRF). Collected variables include demographic information, medical history, risk factors (especially smoking), tumor histology and molecular characteristics (e.g., EGFR, ALK, PD-L1, KRAS, ROS1, RET), ECOG performance status, and treatment modalities across different therapeutic lines.

The registry will also assess real-world treatment patterns and clinical outcomes, including objective response rate (based on RECIST 1.1), progression-free survival (PFS), time to treatment discontinuation (TTD), and overall survival (OS). Adverse events and treatment-related toxicities will be documented and classified according to international standards (CTCAE). A minimum of 1,500 patients per year is expected, with at least 12 months of follow-up per patient.

This project aims to create a reliable national database to support health policy, optimize therapeutic strategies, and guide clinical research. By accounting for variations in clinical practices and patient profiles across the country, SAFRO 2202 is expected to generate robust evidence to improve lung cancer care in Algeria.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed diagnosis of lung cancer (NSCLC, SCLC, or carcinoid tumor)
* Diagnosed at the time of inclusion or within the 12 previous months
* Fully managed (diagnosis, treatment, and follow-up) in an oncology or pulmonology department of one of the 21 participating public/university hospitals
* Signed informed consent obtained

Exclusion Criteria:

* Prior enrollment in this study
* Participation in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with lung cancer (NSCLC, SCLC, or carcinoid tumors), recruited across 21 public or university hospitals in Algeria. Patients must have been diagnosed within 12 months prior to inclusion and be managed entirely within the public healthcare system.
Sampling Method: Non-Probability Sample
Enrollment: 3750 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic and clinical characteristics of lung cancer patients in Algeria | At baseline (inclusion)
  Patient age, sex, smoking history, comorbidities (e.g., COPD, diabetes, cardiovascular disease) and ECOG performance status, collected via eCRFs at inclusion in 21 oncology and pulmonology centers.
Histological type and stage of lung cancer at diagnosis | At baseline (diagnosis/inclusion)
  Histological subtypes (NSCLC, SCLC, carcinoid tumors) and TNM stage of disease at diagnosis.
Molecular profile of tumors | At baseline (inclusion)
  Frequency of molecular alterations (EGFR, ALK, KRAS, PD-L1, ROS1, RET, HER2, NTRK1, BRAF, MET, PIK3CA, MEK1) identified in tumor samples at diagnosis.
First-line treatment modalities | At baseline (initiation of treatment)
  Type of initial treatment received (surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy).

SECONDARY OUTCOMES:
Treatment-related toxicity according to CTCAE | From treatment initiation up to 12 months
  Incidence, type, classification, severity, and impact of adverse events related to lung cancer treatments, assessed with CTCAE criteria.
Objective Response Rate (ORR) | From treatment initiation up to 12 months
  Proportion of patients achieving complete or partial tumor response, assessed according to RECIST 1.1 criteria, based on real-world clinical and radiological data.
Progression-Free Survival (PFS) | From treatment initiation up to 12 months
  Time from treatment initiation to first documented disease progression or death from any cause, whichever occurs first.
Time to Treatment Discontinuation (TTD) | From treatment initiation up to 12 months
  Time from treatment initiation to discontinuation of therapy for any reason, including toxicity, disease progression, or patient/physician decision.
Overall Survival (OS) | Minimum 12-month follow-up after diagnosis
  Time from date of diagnosis to death from any cause, based on real-world clinical follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Adda BOUNEDJAR, Professor of Medical Oncology, Principal Investigator — Frantz Fanon University Hospital, Cancer Center (CAC), Blida, Algeria
Locations (21):
- Algeria (21):
  - Centre Pierre et Marie Curie, Algiers, Algiers Province
  - Chu Beni Messous - Isaad Hassani, Algiers, Algiers Province
  - CHU Mohamed Lamine Debaghine - Bab-el-Oued, Algiers, Algiers Province
  - Chu-Beni Messous - Isaad Hassani, Algiers, Algiers Province
  - EPH Rouiba, Algiers, Algiers Province
  - CLCC Annaba, Annaba, Annaba
  - CLCC Batna, Batna City, Batna
  - CAC-CHU Frantz Fanon, Blida, Blida Province
  - CHU- Hôpital Khelil Amrane, Béjaïa, Béjaia Province
  - CHU Dr Abdesselam Benbadis, Constantine, Constantine Province
  - EH Didouche Mourad, Constantine, Constantine Province
  - CLCC Draâ Ben Khedda, Tizi Ouzou, Draâ Ben Khedda
  - CAC-Laghouat, Laghouat, Laghouat Province
  - CAC Oran EL HASSI- EMIR ABDELKADER, Oran, Oran Province
  - CHU Dr. Benaouda Benzerdjeb, Oran, Oran Province
  - EHS 1er novembre, Oran, Oran Province
  - CAC- Ouargla, Ouargla, Ouargla Province
  - CAC El OUED, El Oued, Oued Souf
  - CAC- Sidi Bel Abbès, Sidi Bel Abbes, Sidi Bel Abbès Province
  - EPH- Sidi Ghiles, Tipasa, Sidi Ghiles
  - CAC-Sétif, Sétif, Sétif Province

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with external researchers. The data will be used exclusively by the study team for the purpose of scientific analysis and publication. No external access to individual-level data is planned.